CLINICAL TRIAL: NCT05336877
Title: Aveir Single-Chamber Leadless Pacemaker Coverage With Evidence Development (ACED) Post-Approval Study
Brief Title: Aveir VR Coverage With Evidence Development Post-Approval Study
Acronym: CED
Status: Recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10426
Record Dates: First submitted 2022-04-11; First posted 2022-04-20 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Cardiac Pacemaker; Arrythmia; Bradycardia
MeSH Terms: conditions — Arrhythmias, Cardiac; Bradycardia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Device: Aveir VR Leadless Pacemaker System: This study will utilize real-world data from patients implanted with the Aveir VR Leadless Pacemaker System. No device intervention is required in this study.
  Interventions: Device: Aveir VR Leadless Pacemaker System
- Device: Single-Chamber Transvenous Pacemaker: This study will utilize real-world data from patients implanted with a single-chamber transvenous pacemaker as a comparator to the Aveir VR LP system study arm. No device intervention is required in this study.
  Interventions: Device: Single-Chamber Transvenous Pacemaker

INTERVENTIONS:
Device: Aveir VR Leadless Pacemaker System — This study will utilize real-world data from patients implanted with the Aveir VR Leadless Pacemaker System. No device intervention is required in this study.
  Groups: Device: Aveir VR Leadless Pacemaker System
Device: Single-Chamber Transvenous Pacemaker — This study will utilize real-world data from patients implanted with a single-chamber transvenous pacemaker as a comparator to the Aveir VR LP system study arm. No device intervention is required in this study.
  Groups: Device: Single-Chamber Transvenous Pacemaker

SUMMARY:
The purpose of this coverage with evidence development (CED) study is to evaluate complications and long-term health outcomes of the single-chamber Aveir Single-Chamber Leadless Pacemaker device (Aveir VR LP).

DETAILED DESCRIPTION:
This is a non-randomized, multi-center study leveraging real-world evidence methods that merge multiple real-world datasets from Abbott and the Center for Medicare Services to compare Aveir VR LP safety and health outcomes to those in patients implanted with single-chamber transvenous pacemakers in a large patient population.

The study will enroll all Medicare patients implanted with the Aveir VR LP and, as the control group, patients implanted with a single-chamber ventricular transvenous pacemaker from any manufacturer.

ELIGIBILITY:
The study cohort will include all Medicare patients with continuous claims data implanted with an Aveir VR leadless pacemaker or a full-system single-chamber ventricular transvenous pacemaker (from any manufacturer) in any US location

Inclusion Criteria:

Medicare beneficiaries implanted with an Aveir VR leadless pacemaker on or after the study start date (i.e., the date of Aveir VR market approval) will be included in the study.

OR

Medicare beneficiaries implanted with a full system (e.g. lead and generator) single-chamber ventricular transvenous pacemaker on or after the study start date

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study cohort will include all Medicare patients with continuous claims data implanted with an Aveir VR leadless pacemaker or a full-system single-chamber ventricular transvenous pacemaker (from any manufacturer) in any US location
Sampling Method: Non-Probability Sample
Enrollment: 8744 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects with Acute Device-Related Complications | 30 days
  Rate of acute complications in subjects implanted with an Aveir VR LP compared to subjects implanted with a single-chamber ventricular transvenous pacemaker. Acute complications are defined as a peri-procedural, device-related adverse event within 30 days post-implant.
Number of Subjects Alive after 2 Years | 2 years
  The 2-year survival rate of subjects implanted with an Aveir VR LP compared with subjects implanted with single-chamber ventricular transvenous pacemaker.

SECONDARY OUTCOMES:
Number of Subjects with Chronic Device-Related Complications | 6 months
  Rate of chronic complications in subjects implanted with Aveir VR LP compared with subjects implanted with a single-chamber ventricular transvenous pacemaker, from 31 days through six months post implant procedure. A chronic complication is defined as a post-procedural, device-related adverse event that requires invasive intervention to resolve.
Number of Subjects with a Device-Related Re-Intervention | 2 years
  Rate of device-related re-intervention in subjects implanted with an Aveir VR LP compared to subjects implanted with a single-chamber ventricular transvenous pacemaker, through 2 years post implant procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Harbert, Study Director — Abbott
Locations (1):
- Abbott, Sylmar, California, United States

IPD SHARING:
Plan to Share IPD: No